CLINICAL TRIAL: NCT04232098
Title: Effect of Feet and Calf Heating on Glucose Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jeff Moore, Primary Investigator, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FEETHEAT
Record Dates: First submitted 2020-01-11; First posted 2020-01-18 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Postprandial Hyperglycemia; Heart Rate Variability
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thermoneutral (No Intervention): thermoneutral condition
- Feet heated (Experimental): Hot water up to ankles
  Interventions: Other: Heat to ankle
- Calf heated (Experimental): Hot water up to top of calves
  Interventions: Other: Heat to calf

INTERVENTIONS:
Other: Heat to ankle — Heat administered via hot water to ankle level
  Arms: Feet heated
Other: Heat to calf — Heat administered via hot water to calf level
  Arms: Calf heated

SUMMARY:
Determine the effect of feet and calf heating on glucose tolerance relative to thermoneutral control. Heat will be administered using hot water (40 degrees celsius).

ELIGIBILITY:
Inclusion Criteria:

* Anyone within specified age range

Exclusion Criteria:

* Anyone outside specified age range

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 30 minute
Blood Glucose | 60 minute
Blood Glucose | 90 minute
Blood Glucose | 120 minute

SECONDARY OUTCOMES:
Blood Pressure | 30 min
Blood Pressure | 60 min
Blood Pressure | 90 min
Blood Pressure | 120 min
Tympanic Temperature | 30 min
Tympanic Temperature | 60 min
Tympanic Temperature | 90 min
Tympanic Temperature | 120 min

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No